CLINICAL TRIAL: NCT00975754
Title: A Phase I, Randomized, Open-label, 5-way Crossover, Single Centre Study in Healthy Subjects to Assess the Lung Deposition of Inhaled Budesonide Delivered Via Different Inhalation Devices
Brief Title: Lung Deposition Via Different Inhalation Devices
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD Carin Jorup, MD, Emerging respiratory, AstraZeneca R&D Lund
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5252M00001
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Healthy Volunteers
Keywords: Inhalation; lung deposition
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Pulmicort pMDI
  Interventions: Drug: Pulmicort pMDI HFA
- 2 (Experimental): Budesonide pMDI
  Interventions: Drug: Budesonide pMDI HFA
- 3 (Experimental): Budesonide pMDI + Aerochamber Zero-stat spacer
  Interventions: Drug: Budesonide pMDI HFA
- 4 (Experimental): Pulmicort repulses via Spira Nebuliser
  Interventions: Drug: Pulmicort Repulses
- 5 (Experimental): Pulmicort Turbohaler
  Interventions: Drug: Pulmicort Turbohaler

INTERVENTIONS:
Drug: Pulmicort pMDI HFA — Inhalation aerosol, 200 μg/ metered dose. Each subject receive a single dose from 4 inhalations
  Arms: 1
Drug: Budesonide pMDI HFA — Inhalation aerosol, 160 μg/ metered dose. Each subject receive a single dose from 4 inhalations
  Arms: 2; 3
Drug: Pulmicort Repulses — Suspension for nebulisation, 0.5 mg/mL. Each subject receive a single dose from 100 inhalations
  Arms: 4
Drug: Pulmicort Turbohaler — Inhaled powder, 200 μg/ metered dose. Each subject receive a single dose from 4 inhalations
  Arms: 5

SUMMARY:
The purpose of this study is to assess the deposition of budesonide to the lung after inhalation with 5 different devices and to relate the findings to in vitro properties of inhaled budesonide.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* BMI between 18 and 30 kg/m2
* Non-smokers/non-snuffers

Exclusion Criteria:

* Pregnant and/or lactating women
* Use of oral contraceptives or hormonal implants
* Known or suspected hypersensitivity to glucocorticosteroids, inhaled lactose, or other excipients in study drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-09; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Lung deposition of budesonide (AUC) | Before dose and repeatadly during the 8-hour period after dose

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, Study Director — AstraZeneca R&D Lund, Sweden; Pia Lena Berg, Principal Investigator — Clinical Pharmacology Unit, AstraZeneca R&D Lund, Sweden
Locations (1):
- Research Site, Lund, Sweden